CLINICAL TRIAL: NCT05291468
Title: PHENOtype Based Therapy With Antibiotics in SARcoidosis Patients With and Without Presence of Cutibacterium Acnes in Granulomatous Tissue
Brief Title: the PHENOSAR Trial: Use of Antibiotics in Treatment of Sarcoidosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Marcel Veltkamp, MD,PhD, Pulmonologist, Principle Investigator, member of staff ILD Center of Excllence, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL73729.100.21
Record Dates: First submitted 2022-02-25; First posted 2022-03-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sarcoidosis, Pulmonary; Sarcoidosis Skin
Keywords: Cutibacterium acnes; antibiotics; azithromycin; doxycycline
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: The study population will be divided in 4 groups Group A consists of patients with C. Acnes present in their tissue Group B consists of patients without C. Acnes present in their tissue 50% of patients in each group will be treated with antibiotics and 50% with placebo.
  Study duration is 4 months
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- C Acnes present in granulomatous tissue, treatment with antibiotics (Active Comparator): patients who are in this arm will receive azithromycin and doxycycline for 3 months
  Interventions: Radiation: FDG-PET/CT
- C Acnes present in granulomatous tissue, treatment with placebo (Placebo Comparator): patients who are in this arm will receive placebo for 3 months
  Interventions: Radiation: FDG-PET/CT
- C Acnes NOT present in granulomatous tissue, treatment with antibiotics (Active Comparator): patients who are in this arm will receive azithromycin and doxycycline for 3 months
  Interventions: Radiation: FDG-PET/CT
- C. Acnes NOT present in granulomatous tissue, treatment with placebo (Placebo Comparator): patients who are in this arm will receive placebo for 3 months
  Interventions: Radiation: FDG-PET/CT

INTERVENTIONS:
Radiation: FDG-PET/CT — Patients will be randomized in a 1:1 ratio to either receive a combination of doxycycline and azithromycin or placebo during 3 months, after which the inflammatory state of disease is measured by FDG-PET/CT and serum biomarkers. If patients have cutaneous sarcoidosis, a skin biopsy will be performed at baseline and at the end of the study.
  Other Names: serum biomarkers; additional skin biopsy

SUMMARY:
In this study it is investigated whether treatment with azithromycin in combination with doxycycline reduces the bacterial load of C. acnes in granulomatous tissue of patients with sarcoidosis and subsequently decreases the inflammatory activation measured by FDG uptake and serum biomarkers.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystemic disease with unknown origin mostly affecting intrathoracic lymph nodes, lungs and skin. Sarcoidosis is characterized by the formation of non-caseating granulomas causing a variety of symptoms based on the organs involved. Although frequently described as a benign disease, mortality rate has been estimated to be around 11.0 per 1000 person-years in patients with sarcoidosis, with respiratory failure as the most common cause of death in the western world.

The main treatment indication in sarcoidosis is risk of organ failure. In the literature the need for systemic treatment varies between 20-70%. Since there is no curative treatment for sarcoidosis, treatment is focused on suppression of the inflammation. This is usually done with the use of immunosuppressive drugs, such as prednisone and/or methotrexate, and in patients with severe refractory disease infliximab. It is well known that treatment with immunosuppressive drugs is associated with burdensome side effects for patients and impaired quality of life.

Considerable research has been done on the possible role C. acnes in the pathogenesis of sarcoidosis. In a recent work of our own group it was shown that presence of C. acnes within granulomatous tissue can be detected in 41% of Dutch patients with sarcoidosis. Azithromycin has an inhibiting effect on several bacterial infections, such as C. acnes. Therefore, sarcoidosis patients with C. acnes in the granulomatous tissue might benefit from treatment with azithromycin. Given the fact that microbial resistance to azithromycin is relatively easy to develop, it is common practice to treat C. acnes with a combination of azithromycin and doxycycline.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis.
* No treatment indication for the sarcoidosis
* Inflammatory activity according to FDG-PET scan at baseline
* SUVmax above 3 in the lung and/or above 5 in mediastinum/hili

Exclusion Criteria:

* Increased duration of QT interval (>440ms for men and >450ms for women) on ECG
* Hearing deficits, as this is a possible side effect of azithromycin
* Being pregnant or breastfeeding at time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 2 weeks
  Difference of standarized uptake value (SUVmax) uptake after treatment with antibiotics between patients with and without C. acnes in their granuloma

SECONDARY OUTCOMES:
lung function | 2 weeks
  Difference in FVC after treatment with antibiotics between patients with and without C. acnes in their granulomatous tissue
quality of life according to questionnaire | 2 weeks
  Monitor quality of life for patients treated with antibiotics compared to patients receiving placebo, measured by King's Sarcoidosis Questionnaire that is taken at baseline and end of study. QOL is measured with the King's Sarcoidosis Questionnaire (KSQ), which is a validated questionnare on sarcoidosis with 5 scales and 29 items.

OTHER OUTCOMES:
serum biomarker: ACE | 2 weeks
  Determine whether treatment with azithromycin and doxycycline changes levels of serum biomarker Angiotensin Converting Enzyme (ACE) in U/I in sarcoidosis patients
serum biomarker: IL-2R | 2 weeks
  Determine whether treatment with azithromycin and doxycycline changes levels of serum biomarker interleukin-2receptro (IL-2R) in pg/mL in sarcoidosis patients

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No
data of patients will be coded and will not be traceable to a specific participant when used by other researchers